CLINICAL TRIAL: NCT01005186
Title: Changing Lifestyle in Children: All Change: Can This Reduce Cardiovascular Risk?
Brief Title: Changing Lifestyle in Children
Acronym: ALLChange
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: University of St Andrews (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2003CV40
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Risk
MeSH Terms: interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Active
  Interventions: Behavioral: Eating habits, diet and exercise
- Active 2 (Experimental): Active
  Interventions: Behavioral: Eating habits, diet and exercise

INTERVENTIONS:
Behavioral: Eating habits, diet and exercise — Programme of change to eating habits, diet and exercise

SUMMARY:
A lifestyle intervention aimed at improving exercise levels in primary school children.

ELIGIBILITY:
Inclusion Criteria

* Children 9-11 yrs

Exclusion Criteria:

* Children <9 yrs and >12 yrs

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2006-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Can an acceptable strategy, based on social cultural factors that influence adherence to the strategy and designed for altering lifestyle associated with CV risk (ALL CHANGE) be developed for school aged children?

SECONDARY OUTCOMES:
Is ALL CHANGE more effective in altering lifestyle than conventional health education delivered as part of the school curriculum?